CLINICAL TRIAL: NCT02709226
Title: A Phase I Dose Escalation Trial of Re-Irradiation in Good Prognosis Recurrent Glioblastoma
Brief Title: Dose Escalation Trial of Re-irradiation in Good Prognosis Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 160081; 16-C-0081
Record Dates: First submitted 2016-03-15; First posted 2016-03-16 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-16

CONDITIONS: Astrocytoma, Grade IV; Giant Cell Glioblastoma; Glioblastoma Multiforme; Gliosarcoma
Keywords: Brain Tumor; Astrocytoma; GBM; Radiation Therapy
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Astrocytoma | interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/Radiation (Experimental): Dose escalation is as follows: dose level 1 (DL1) 3.5 Gy x 10; dose level 2 (DL2) 3.5 Gy x 12; dose level 3 (DL3) 3.5 Gy x 14. If 2 DLTs are observed in the second dose level a step down dose of 3.0 Gy x 14 fractions will be tested. If 2 DLTs are observed in the third dose level a step down dose of 3.0 Gy x 17 fractions will be tested. The study will have 3 planned re-irradiation dose levels, with 1 to 6 patients per dose level using the 3+3 design to define the MTD. The number of patients may be increased to 9 total patients at the MTD ( provided no DLT) with a maximum of 21 evaluable patients enrolled.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation therapy will be administered daily Monday-Friday at NCI, ROB unless the treatment schedule requires amendment in the event of inclement weather or federal holidays. Radiation therapy dose will be administered as per on consecutive treatment days, 5 fractions per week via a linear accelerator using 6 MV photons or greater. Dose escalation is as follows: dose level 1 (DL1) 3.5 Gy x 10; dose level 2 (DL2) 3.5 Gy x 12; dose level 3 (DL3) 3.5 Gy x 14. If 2 DLTs are observed in the second dose level a step down dose of 3.0 Gy x 14 fractions will be tested. If 2 DLTs are observed in the third dose level a step down dose of 3.0 Gy x 17 fractions will be tested. The study will have 3 planned re-irradiation dose levels, with 1 to 6 patients per dose level using the 3+3 design to define the MTD. The number of patients may be increased to 9 total patients at the MTD ( provided no DLT) with a maximum of 21 evaluable patients enrolled.

SUMMARY:
Background:

A glioblastoma is a tumor in the brain. It is treated with surgery, chemotherapy and radiation therapy. However, most people s tumors come back after therapy. When the tumor grows back, surgery or chemotherapy may not be possible or may no longer work. Repeat radiation therapy or re-irradiation, is an option for treating these tumors when they regrow.

Objective:

To find out the safety and highest tolerated dose of re-irradiation for people who have recurrent glioblastoma.

Eligibility:

People ages 18 50 who have glioblastoma that has been treated with radiation but has regrown.

Design:

Participants will be screened with:

Medical history

Physical exam

MRI of the brain: They will lie in a machine that takes pictures of the brain.

Participants will have baseline tests before they start therapy. These will include:

Blood tests

Neuropsychological tests: These test things like memory, attention, and thinking.

Quality of life questionnaire

Eye and hearing tests

Participants will get a CT of the brain prior to radiation start in order to plan the radiation treatment. Once the plan is completed, they will receive radiation once a day Monday Friday for a total of 10 17 treatments. They will lie on their back for about 10 minutes while they get the treatment.

Participants will be monitored for side effects.

After they finish treatment, participants will have visits 1, 2, and 3 months later. Then they will have them every 2 months for 3 years. These will include:

Medical history

Physical exam

Blood tests

MRI of the brain.

Quality of life questionnaire

Neuropsychological tests (at some visits)

After 3 years, participants will be contacted by phone each month.

DETAILED DESCRIPTION:
Background

* Although the survival of gliomas has improved, most high grade gliomas will recur in field or adjacent to the treatment field within months to years of the original treatment. In newly diagnosed GBM, the concurrent use of radiation and temozolomide is standard of care.
* Surgical resection upon recurrence is possible in less than 50% of patients. For a significant proportion of recurrent glioma patients in whom reresection is not favourable and for whom systemic options have been exhausted, re-irradiation has emerged as a possible treatment option.
* Using modern precision RT techniques (stereotactic radiosurgery (SRS), stereotactic radiotherapy (SRT) or intensity modulated radiation therapy (IMRT), Rapid Arc techniques), re-irradiation has proven a feasible option with possible benefit in outcome as these techniques are often able to minimize dose to previously treated organs at risk in the field (OAR) and treat the recurrence safely.
* Data from multiple retrospective studies has indicated that not only is re-irradiation feasible, but it may actually improve survival in the appropriately selected patient.

Objective

The primary objective of this phase I study is to determine maximum tolerated re-irradiation dose (MTD).

Eligibility

* Recurrent glioblastoma or gliosarcoma
* Prior standard radiation therapy to a dose ranging from 50 to 60 Gy at 1.8 to 2 Gy per fraction.
* Prior irradiation > 12 months from enrollment on protocol.
* Age greater than or equal to 18.
* KPS greater than or equal to 70

Design

* Radiation therapy will be administered daily Monday-Friday at Radiation Oncology Branch (ROB), NCI. All the protocol related follow-up appointments will occur at NCI ROB. Radiation therapy dose will be administered on consecutive treatment days, 5 fractions per week via a linear accelerator using 6 MV photons or greater. Using a 3 plus 3 design , and three dose escalation levels, with 6 patients per dose level with 9 total patients at the MTD (provided no DLT), a maximum of 21 evaluable patients will be enrolled.
* Time to progression will be determined by the interval from initiation of treatment on protocol to progression as per RANO criteria.
* Neurologic decline without radiographic evidence of tumor will be designated as treatment related toxicity. Survival duration will be determined by the interval from initiation of treatment on protocol to date of death.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Histological diagnosis

     Previous histologic diagnosis of glioblastoma, transformation to glioblastoma or gliosarcoma established by biopsy or resection prior to enrollment as evident on NIH or outside pathology.
  2. Patients must be age greater than or equal to 18.
  3. Patients should have a KPS greater than or equal to 70%
  4. Prior standard radiation therapy to a dose ranging from 50 to 60 Gy at 1.8 to 2 Gy per fraction.
  5. Patients must be more than or equal to 14 days from previous cytotoxic treatment.
  6. Concurrent therapy

     The concurrent use of bevacizumab is allowed if previously initiated for tumor progression or symptomatic management. Prior temozolomide or other cytotoxic chemotherapy is allowed.
  7. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
  8. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

1. Prior therapy < than 2 weeks since surgical re-resection or biopsy
2. Pregnant or breast feeding females are excluded due to potential mutagenic effects on the developing fetus or newborn
3. Preexisting grade 3 or 4 nervous system disorder as per CTCAE Version 4.0
4. Clinically significant unrelated systemic illness (including but not limited to active life threatening infection, cardiac or neurologic events, current hospital admission for a coexisting comorbid illness), which would make it impossible for the patient to tolerate re-irradiation or systemic chemotherapy or likely to interfere with the results.
5. Patients exhibiting baseline grade 3 or 4 by CTCAE criteria are excluded due to difficulty in assigning these to the study intervention as treatment related DLT.
6. Patients with preexisting known or suspected radiation sensitivity syndromes will be excluded due to potential confounding effect on outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
To determine maximum tolerated re-irradiation dose (MTD). | 1 month after completion of re-irradiation
  The MTD will be based on the assessment of DLT within one month following the re-irradiation, and will be defined as the dose level at which less than one-third of patients (0/3 or 0-1/6 patients) treated at that dose experience a DLT, with the next higher dose level demonstrating a one-third or greater number of patients (>= 2/3 or >= 2/6 patients) having DLT.

SECONDARY OUTCOMES:
To determine QOL and impact on neurocognition in the setting of re-irradiation of recurrent glioblastoma | baseline and at each visit
  QOL scores will be summarized at baseline and for each visit. Changes from baseline of health-related quality of life questionnaire mean scores will be evaluated
To determine progression free survival and overall survival. | time of progression; time of death
  interval from initiation of treatment on protocol to progression as per RANO criteria Survival duration will be determined by the interval from initiation of treatment on protocol to date of death
To determine late toxicity secondary to re-irradiation | completion of study
  listing of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0081.html